CLINICAL TRIAL: NCT00898742
Title: Molecular Signatures of HNSCC in Response to Targeted Therapies
Brief Title: Gene and Protein Expression Patterns in Predicting Response to Cetuximab in Patients With Recurrent and/or Metastatic Head and Neck Cancer
Status: Terminated | Type: Observational
Why Stopped: study closed prematurely upon PI's departure from VICC
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Murphy, MD, Professor of Medicine, Medical Oncologist, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC HN 0715; P30CA068485 (NIH); VU-VICC-HN-0715; VU-VICC-070668
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2013-03

CONDITIONS: Head and Neck Cancer
Keywords: recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent verrucous carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; recurrent squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; salivary gland squamous cell carcinoma; stage IV salivary gland cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Salivary Gland Neoplasms | interventions — DNA; Tissue Array Analysis; Reverse Transcriptase Polymerase Chain Reaction; Mass Spectrometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- head and neck cancer patients
  Interventions: Genetic: DNA and tissue microarray analysis; Genetic: reverse transcriptase-polymerase chain reaction; Other: mass spectrometry

INTERVENTIONS:
Genetic: DNA and tissue microarray analysis — The lab has a candidate gene expression signature for the prediction of the cetuximab response. It may be possible to identify patients who will respond to cetuximab based on the patterns of gene and protein expression.
Genetic: reverse transcriptase-polymerase chain reaction — The lab has a candidate gene expression signature for the prediction of the cetuximab response. It may be possible to identify patients who will respond to cetuximab based on the patterns of gene and protein expression.
Other: mass spectrometry — The lab has a candidate gene expression signature for the prediction of the cetuximab response. It may be possible to identify patients who will respond to cetuximab based on the patterns of gene and protein expression.

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how will patients respond to treatment.

PURPOSE: This research study is looking at gene and protein expression patterns in predicting response to cetuximab in patients with recurrent and/or metastatic head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify 100 patients from the Head and Neck Tumor Tissue Repository and Clinical Database treated with cetuximab monotherapy or cetuximab-containing combination therapy as a standard of care for recurrent and/or metastatic head and neck squamous cell carcinoma at Vanderbilt University Medical Center.
* To assay the diversity of gene and protein expression patterns seen in these patients.
* To identify predictive patterns associated with treatment response and survival of these patients by correlating the laboratory data with clinical data.

OUTLINE: Tumor tissue specimens and clinical data are obtained from the Head and Neck Tumor Tissue Repository and Clinical Database protocol VU-VICC-HN-0356. Specimens are analyzed for patterns of gene and protein expression predictive of cetuximab treatment response and survival by DNA microarray, tissue microarray, reverse transcriptase-PCR, and mass spectroscopy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of recurrent and/or metastatic head and neck squamous cell carcinoma

  * Enrolled on the Head and Neck Tissue Repository and Clinical Database protocol VU-VICC-HN-0356
  * Previously treated with cetuximab monotherapy or cetuximab-based combination therapy
* Sufficient biological material available for analysis

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: head and neck cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2007-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Identification of 100 patients from the Head and Neck (H&N) Tumor Tissue Repository and Clinical Database treated with cetuximab or cetuximab-containing combination therapy as a standard of care | approximately three years from enrollment of first patient
Gene and protein expression patterns in selected H&N Tumor Tissue Repository and Clinical Database patients | upon colleciton of final patient data
Predictive patterns of gene and protein expression associated with cetuximab treatment response and survival | upon collection of final patient data

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Murphy, MD, Study Chair — Vanderbilt-Ingram Cancer Center
Locations (3):
- United States (3):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center at Franklin, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee